CLINICAL TRIAL: NCT06755931
Title: The Effect of Quilling Exercise Applied Before Cardiac Catheterization and Angiography on Fear and Anxiety in Children: Randomized Controlled Study
Brief Title: The Effect of Quilling Exercise Applied Before Cardiac Catheterization and Angiography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semra Kose (Other)
Responsible Party: Sponsor-Investigator, Semra Kose, Assistant Professor (PhD, RN), Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NEU2024YLTez(2)
Record Dates: First submitted 2024-12-15; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Children; Cardiac Catheterization
Keywords: child; Cardiac catheterization; fear; anxiety; nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study was planned as a pre-test, post-test parallel group (intervention-control), randomized controlled experimental research type.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quilling Group (Experimental)
  Interventions: Behavioral: quilling set
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: quilling set — After the intervention group is determined in randomization, half an hour before the cardiac catheterization and angiography procedure, without premedication treatment, the researcher will be asked to choose 2 animal and plant figures, samples of which have been previously made, through a quilling set, in cooperation with the researcher. It will be done with the child in a 15-20 minute period, accompanied by the researcher, with 2 figures chosen by the child. With the opportunity for the child to choose the color and figure he/she wants, the child will be at the center of the work. The figure will be given as a gift to the child and the survey forms will be filled out again 5 minutes after the application, before the premedication treatment. In order to prevent bias in the research, the descriptive information form and fear and anxiety scales will be taken by the evaluation of three people: the researcher, the parent and the child.
  Arms: Quilling Group
Behavioral: Control — Before the procedure, while the child is in the patient room, the details of the research will be explained, their consent will be obtained and the Introductory Information Form will be filled in by the parent, and the Fear Scale and State Anxiety Scale will be filled in by the child and the parent. After the control group is determined in randomization, the researcher will apply the posttest without premedication treatment half an hour before the cardiac catheterization and angiography procedure. No separate intervention will be applied. In accordance with ethical principles, after the procedure, 2 Quilling figures chosen by the control group and the child will be prepared with the help of the researcher, and the prepared figures will be gifted to the child.
  Arms: Control

SUMMARY:
The heart is one of the most important organs of the body. Any defect in the heart or blood vessels can cause serious problems and include a number of health problems that reduce the quality of life. Despite recently developing technologies, heart diseases are one of the important causes of morbidity and mortality in children. He contributed to the determination of the treatment plan in more than 84% of the cases in cardiac catheterization and angiography, which are widely used in the diagnosis and treatment of congenital heart diseases. Since the cardiac catheterization and angiography procedure consists of a process, the nurse plays an important role in shortening the treatment time, increasing the comfort level, and reducing anxiety and fear as a result of the correct interventions that follow the patient before, during and after the procedure. For this reason, the nurse must be equipped and have sufficient knowledge in the field in the nursing care and interventions applied to patients for whom angiography is planned. Since cardiac catheterization and angiography is an invasive procedure and requires surgical intervention, it can cause negative situations such as fear, pain and anxiety in children. Since it is thought that it can be effective in reducing fear and anxiety in children through the Quilling Set activity planned to be implemented in the study in order to reduce the negative situations caused by the procedure, it is thought that the study will make a positive contribution to children and parents in physical and psychological terms.

DETAILED DESCRIPTION:
Cardiac catheterization and angiography is an invasive interventional cardiology method that helps diagnose coronary artery diseases by revealing the anatomy, physiology and pathophysiology of the heart and circulation. It can be performed for diagnosis and treatment purposes. Although the usefulness of diagnostic cardiac catheterization in the clinical setting has diminished in recent years with the advent of non-invasive imaging modalities such as echocardiography, magnetic resonance imaging, and computed tomography, diagnostic catheterization is still a valuable tool in the evaluation of pediatric heart disease. Cardiac catheterization and angiography are preferred over noninvasive methods in cases where it is important to precisely determine the disease anatomy (pulmonary atresia, fallot tetralogy, etc.). Since the procedure can typically be performed with minimal invasion, its use is common in pediatric patients. In addition to the presence of chronic disease in children, the fear of hospitalization and surgical operation for cardiac catheterization and angiography constitutes a serious source of stress. Studies show that children experience pain, anxiety, fear and stress during these medical procedures. These fears are a cause for anxiety for both the child and the family. In addition, the experience directly affects the child's hospital process, treatment and care experience in the future, so it is of great importance to control fear and anxiety in children. For a child and parent with a chronic disease, returning to the hospital causes the child to fear and feel anxious about factors such as illness and medication. For this reason, not only a child-centered approach but also a family-centered holistic nursing approach should be followed in the nursing care of a child with a chronic disease. It is reported in the literature that children with congenital heart disease experience physical, emotional, behavioral and neurodevelopmental problems. The process of chronic heart disease includes accepting the existing situation, tolerating difficulties, and making life easier by arranging daily activities. Since the cardiac catheterization and angiography process consists of a process, the nurse plays an important role in shortening the treatment time and increasing the comfort level as a result of the correct interventions that follow the patient before, during and after the procedure. The nurse, who is with the child at almost every stage of the procedure, is in an important position to monitor and manage the children's fear, anxiety and pain symptoms.

In recent years, nursing research has focused on the management and reduction of procedural pain in children and the use of non-pharmacological methods to relieve anxiety and stress. The most common of these methods are massage, distraction, positioning, and watching videos. For example, Karakul et al. It reveals that musical intervention applied during pediatric cardiac catheterization in children affects the reduction of pain, fear and anxiety levels and the stabilization of vital signs.

Kim et al. According to a study conducted by Kim et al., it was observed that hearing the recorded mother's voice reduced anxiety, agitation on awakening, and the need for anesthesia in children undergoing cardiac catheterization and angiography. Agüero et al. suggested that short-term interventions performed by nurses before urological surgery in children could reduce preoperative anxiety. Wang et al. It has been suggested that music and animation strategies can significantly reduce anxiety in children before tonsillectomy or adenoidectomy surgery and improve surgical cooperation during anesthesia induction.

As a result, when the literature was scanned, it was determined that cardiac catheterization and angiography caused fear and anxiety in children because they were invasive procedures, and it was seen that additional non-pharmacological studies were needed to reduce fear and anxiety in children. The aim of the study was to evaluate the effect of the Quilling set on fear and anxiety in children as it could be a new non-pharmacological intervention, as the Quilling set study to be applied to children with cardiac catheterization and angiography is not included in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 9-12,
* Able to read and write Turkish,
* Accompanied by their parents,
* Having no mental disabilities or communication problems,
* No visual or hearing impairment,
* Those who have not had cardiac catheterization or angiography before,
* Children who are willing to participate in the research will be included in the research.

Exclusion Criteria:

* Those who have any body function deficiency that prevents them from playing quilling,
* Those who did not complete the quilling initiative and wanted to quit the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | During the children's first hospitalization, the researcher will fill out an introductory information form. (Approximately 5 minute)
  In the introductory information form prepared by the researcher in line with the literature; There are a total of 11 questions, such as the child's age, gender, number of siblings, family type, place of residence, family income level, mother's age, mother's education, mother's profession, and hospitalization status of the child.
State Anxiety Inventory for Children (STAI-C) | It will be filled out by the researcher, child and parent before and after the procedure (Approximately 10 minute).
  This scale was developed by Spielberger in 1973 to evaluate children's state and trait anxiety and is in a self-report form. It was translated into Turkish by Özusta and an application study was carried out. As a result of some procedures, the scale was turned into 2 separate scales containing a total of 40 items (20 state and 20 trait anxiety items). Although the validity and reliability of the scale has been done for children aged 9-12, the scale can be used until the age of 17 because it is difficult for children over the age of 12 to understand the adult anxiety scale. It has also been seen in the literature that it is used in all school-age children who can read. In the STAI-C, children are asked to mark one of three options regarding how they feel "at that moment". The scale aims to evaluate emotions related to state anxiety such as tension, irritability, rush, and uneasiness.The highest score that can be obtained from the STAI-C is 60 and and the lowest score is 20.
Child Fear Scale | It will be filled out by the researcher, child and parent before and after the procedure (Approximately 10 minute).
  This scale was used by McMurtry et al. to measure children's anxiety levels. It was developed by in 2011. The scale was developed by Gerçeker et al. in 2018. It has been validated in Turkish by and is aimed at children aged 5-10. However, it is stated that it can be used up to the age of 12. Facial muscle changes in fearful expressions were drawn by a graphic designer based on photographs of frightened faces. The scale can be used by the family, the child or the researcher to evaluate children. In this scale, the child is shown a scale containing five facial expressions rated between 0 and 4 points. While 0 indicates no fear and anxiety; 4 shows the highest fear and anxiety. These are: "0" neutral expression (no anxiety), "1" very little fear (very little anxiety), "2" some fear (some anxiety), "3" more fear (more anxiety), "4" the most fear possible. It is considered high fear (severe anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No